CLINICAL TRIAL: NCT07175532
Title: Prospective Multicenter Registry of Patients With Mitral Stenosis Undergoing Percutaneous Mitral Balloon Commissurotomy
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Min Song, Professor, Asan Medical Center
Other Study IDs: 2025-0396
Record Dates: First submitted 2025-09-15; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the clinical outcomes after percutaneous mitral balloon commissurotomy (PMBC) for patients with mitral stenosis (MS) using nation-wide multicenter prospective registry including tertiary-referral hospitals in Korea.

The main question it aims to answer is:

What is the clinical outcomes after PMBC? Which method is appropriate to determine inflated Inoue balloon size?

ELIGIBILITY:
Inclusion Criteria:

* Patients with mitral stenosis undergoing PMBC

Exclusion Criteria:

* Patients who cannot understand this study due to mental illness
* Serious comorbidity limiting life expectancy within 1 year
* Limited activity (NYHA class III or IV) due to non-cardiac disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mitral stenosis undergoing PMBC
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | From enrollment to 1 year after PMBC

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea